CLINICAL TRIAL: NCT02645292
Title: Comparison Between Stair Climbing and One Mile Walking in Relation to Cardiorespiratory Fitness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Mr, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U/SERC/83/2015
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 mile Walk using treadmill (Experimental): Walking for 1 mile on treadmill (American Motion Fitness, 8800D) as fast as participant can, without any inclination
  Interventions: Device: 1 mile walk using treadmill
- Stair Climbing (Experimental): 30 meters of vertical distance to be covered (14 flights of stairs with a total of 154 steps)
  Interventions: Device: Stair Climbing

INTERVENTIONS:
Device: 1 mile walk using treadmill — Walk for 1 mile on treadmill (American Motion Fitness, 8800D) at self selected speed as fast as participant can without any inclination.
  Arms: 1 mile Walk using treadmill
Device: Stair Climbing — Climb 14 flights of stairs at self selected speed. No double step at a time and running allowed.
  Arms: Stair Climbing

SUMMARY:
The worldwide epidemic of physical inactivity is rising significantly and the main cause is sedentary lifestyle. In this era of globalization and rapid advancement of technology, people are chasing after worldly matters, leading them to abandon the most important factor in their life and that's their body. Most people are leading a sedentary lifestyle as they indulge themselves in their never-ending work. There is a significant lack of awareness on the importance of physical activity and cardiorespiratory fitness to health as people are focusing more on factors such as smoking, cholesterol and hypertension. The purpose of this study is to evaluate the effectiveness of stair climbing (SC) and 1 mile walking (1MW) in relation to cardiorespiratory responses and fitness.

DETAILED DESCRIPTION:
The incidences of chronic diseases and cardiovascular diseases are escalating rapidly and fingers are being pointed to physical inactivity and poor cardiorespiratory fitness as one of the few main 'predictors of premature mortality. According to WHO (2015), 23% of adults above the age of 18 years old were insufficiently physically active in 2010, with men scoring 20% and women 27%. Comparing high income and low income countries, 26% of men and 35% of women of high income countries was said to be insufficiently physically active compared to 12% of men and 24% of women of low income countries. This may be due to the fact that people of high income countries are more engrossed in chasing after worldly matters at work and preferring a sedentary lifestyle at home after work. Globally, adolescents between the age of 11 to 17 years old scored a high percentage of 81% of being insufficiently physically active and this may be because adolescents prefer to spend more time on internet, playing games on computers or watching dramas or movies. In the Physical Activity Statistics 2015 by the British Heart Foundation, it is reported that North West of England has the highest level of physical inactivity with 26% for men and 31% for female. It was also mentioned that household incomes play a role in the level of physical activity in England. In 2012, 29% men and 34% women from the lowest quintile of household income in England were physically inactive compared to 11% men and 18% women of the highest quintile of household income.[1] In Malaysia a research conducted on physical activity index among Malaysian youth and out of 1801 respondents, 23% men and 31.3% women were insufficiently physically active.[2] In another research on the Prevalence and Factors Associated with Physical Inactivity among Malaysian Adults, the overall prevalence of physical inactivity was 43.7%.[3] Similar to other researchers, results also show that women are more physically inactive at 9 465 (50.5%) out of 18 744 female respondents compared to men at 5367 (35.3%) out of 15205 male respondents. It is important to ensure that everyone participates in physical activities in effort to improve their health and indirectly reduce the risk of mortality. Hence, the researcher aims to compare the effects of stair climbing and one mile walking in relation to cardiorespiratory responses and fitness to find which one is better compared to other as these type of activates can be performed in any settings and does not require sophisticated equipments.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary Adults
* Height:160cm to 170cm
* Willing to participate

Exclusion Criteria:

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Physical Fitness Index | At baseline and at end of 4 weeks of intervention
  ''Change'' is being assessed
V02max | At baseline and at end of 4 weeks of intervention
  ''Change'' is being assessed

SECONDARY OUTCOMES:
Recovery Heart Rate | At baseline and at end of 4 weeks of intervention
  ''Change'' is being assessed
Systolic & Diastolic Blood Pressure | At baseline and at end of 4 weeks of intervention
  ''Change'' is being assessed
Respiratory Rate | At baseline and at end of 4 weeks of intervention
  ''Change'' is being assessed
Rate of Perceived Exertion | At baseline and at end of 4 weeks of intervention
  ''Change'' is being assessed

IPD SHARING:
Plan to Share IPD: No
It is confidential

REFERENCES:
- [Background] 1. Townsend N, Wickramasinghe K, Williams J, Bhatnagar P, Rayner M (2015). Physical Activity Statistics 2015. British Heart Foundation:London
- [Background] 2. Salamudin, N., & Harun, M. (2013). Physical Activity Index among Malaysian Youth. Asian Social Science, 9(12).
- [Background] Ying C, Kuay LK, Huey TC, Hock LK, Hamid HA, Omar MA, Ahmad NA, Cheong KC. Prevalence and factors associated with physical inactivity among Malaysian adults. Southeast Asian J Trop Med Public Health. 2014 Mar;45(2):467-80. PMID 24968689